CLINICAL TRIAL: NCT04059809
Title: Photobiomodulation for Breast Cancer Radiodermatitis Prevention. A Randomized Controlled Trial.
Brief Title: Photobiomodulation for Breast Cancer Radiodermatitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AC Camargo Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2.777.676
Record Dates: First submitted 2019-08-13; First posted 2019-08-16 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer; Radiodermatitis; Radiotherapy Side Effect; Radiation Dermatitis; Radiation Toxicity; Radiation Injuries; Quality of Life; Breast Neoplasms
Keywords: Laser; Photobiomodulation; Radiodermatitis; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Radiodermatitis; Radiation Injuries | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Randomized single blind controlled trial
Who Masked: Participant, Care Provider
Masking Description: The participant and care provider will be blinded regarding the status of photobiomodulation device (if switched on or off).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): The control group will have usual care according to the orientation of the radiation therapy faculty responsible for the radiotherapy treatment the PBM device will be switched off
- Photobiomodulation (PBM) (Experimental): Additionally to the usual care, the patients will receive the PBM. Treatment will be done twice a week.
  Interventions: Device: Photobiomodulation

INTERVENTIONS:
Device: Photobiomodulation — Photobiomodulation will be with the Cicatrillux (Cosmedical®) LED that contains 36 red light emitters in a 10x12 cm neoprene plate with 650 nm LED wave length whose optical spot diameter is 5 mm and with an average wave length of 2 ~ 5 mw for 10 minutes that will be placed over the area that will be irradiated for 10 minutes;
  Arms: Photobiomodulation (PBM)

SUMMARY:
A prospective single blind controlled randomized trial to evaluate the superiority of photobiomodulation (PBM) using LED-therapy in reducing the prevalence of radiodermatitis in breast cancer compared to usual local care.

DETAILED DESCRIPTION:
Breast cancer is the second most common cancer in the world, the most common among women in Brazil and accounts for approximately 25% of new cases of cancer in women. One of the pillars of treatment is the radiotherapy, being able to generate a toxic effect in the neoplastic cells and also deleterious in healthy cells, with early and late side effects, being radiodermatitis one of these affections. Moreover, radiodermatitis may cause discontinuation of radiotherapy until the skin is able to receive the appropriate dose. Photobiomodulation (PBM) is a non-invasive, a-thermal treatment modality based on the effect of light in biological systems leading to the activation of epithelial healing through the modulation of several metabolic processes through photochemical reactions. PBM use in an oncologic setting has become an interesting object of study in recent years and even though there are different possibilities for the use in breast cancer and physicians are not yet familiar with this therapy. Several in vitro studies with different cell types ranging from keratinocytes, endothelial cells and fibroblasts have been performed showing that PBM is capable of enhancing cell migration, proliferation, local metabolism, inducing collagen synthesis and secretion of growth factors, self-regulation of the production of proinflammatory cytokines and cellular apoptosis, aiding in the recovery of the dermis and epidermis. The aim of this study will be to evaluate the superiority of the use of photobiomodulation using LED-therapy in relation to the development of radiodermatitis in breast cancer compared to usual local care.

The study will included 110 women after informed consent will be randomly assigned into two groups. There will be 11 groups of 10 envelopes each, where each group will contain a code that allocates patients in group A (05 patients) and group B (05 patients). After the allocation of the 10 patients, a new envelope group will be available until the total number of patients scheduled for this study is reached (110, 55 in each group). Group A (GA) will be the control group of usual care according to the orientation of the radiation therapy clinic responsible for the radiotherapy treatment and with the use of the PBM device switched off. Group B (GB) will be the intervention group, which in addition to the usual care oriented in the radiotherapy clinic responsible for the radiotherapy treatment will use the attached PBM. Both groups will use a pair of glasses that will block the visualization of the light emitted by the PBM device, precisely so that they do not know in which research group it is located. Treatment will be done twice weekly, Tuesday and Thursday. The Photobiomodulation will be with the Cicatrillux (Cosmedical®) LED that contains 36 red light emitters in a 10x12 cm neoprene plate with 650 nm LED wave length whose optical spot diameter is 5 mm and with an average wave length of 2 ~ 5 mw for 10 minutes that will be placed over the area that will be irradiated for 10 minutes; the LED board will be wrapped in a plastic film that will be changed between each use. Both, the control group and the intervention group, will be evaluated for radiodermatitis by the oncologist who accompanies them and by a nurse, and both evaluators will not know in which group the person evaluated belongs. Concomitant to the radiotherapy sessions, both groups will be evaluated by a clinical and sociodemographic questionnaire, by the "Behavioral Risk Factor Surveillance System" (BRFSS), by the Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH) by the Analog Visual Scale for Pain, Radiodermatitis Assessment through the Radiation Therapy Oncology Group (RTOG), application of the European Organization for Research and Treatment of Breast Cancer-Specific Quality of Life Questionnaire questionnaire (EORTC QLQ-BR23) and the European Organization for Research and Treatment of Cancer (EORTC QLQ-30), all questionnaires have already been translated and validated into the Portuguese language. The classification of radiodermatitis and pain assessment will be repeated 90 days after the start of radiotherapy. A descriptive and comparative analysis of the intervention groups will be performed in relation to the selected variables. The evaluation of the outcomes will be performed by intention to treat and by adherence to the protocol, through relative risk, and 95% confidence interval. To analyze the data will be used "Statistical Package for Social Sciences" (SPSS) v.23 Demo (SPSS Inc., Chicago, Illinois, United States). The McNemar test will be used to compare pain levels between groups. For inter-group assessments of the proportion of radiodermatitis, the chi-square test will be used to compare the intervention and control of the group.

Secondary objectives will be to describe the socio-demographic and clinical characteristics of the studied population; to evaluate the incidence of radiodermatitis in people with breast cancer, immediately after and 90 days post-radiotherapy according to study intervention group; to evaluate the adherence and satisfaction to treatment with PMB using LED-therapy in people with breast cancer; to compare the occurrence of pain and its graduation according to the intervention group, immediately after the radiotherapy and in the follow-up of 90 days in people with breast cancer; to evaluate the quality of life of people submitted to radiotherapy for breast cancer according to the intervention group and changes in radiotherapy treatment.

The inclusion criteria are women older than 18 years with histological diagnosis of breast cancer who underwent conservative surgery or mastectomy, without immediate breast reconstruction, treated with conventional radiotherapy referred by the oncologist who accompanies her regularly and who have availability of 20 minutes before the radiotherapy session to CORSB Radiation Therapy and Megavoltage to apply the LED-therapy and accept to participate in the research signing the Free and Informed Consent Term (TCLE). Patients who have undergone mastectomy with immediate breast reconstruction and those who suffer from collagen diseases will be excluded from this study.

The investigators hypothesized that photobiomodulation can stop the progression of radiodermatitis or lead to a faster cure, in turn, would have beneficial effects on the quality of life of these people. Then, it is expected that, at the end of radiotherapy sessions, people treated with therapy would have less severe skin reactions and higher quality of life when compared to people in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer
* Mastectomy or breast conserving surgery
* Informed consent
* Radiotherapy schedule completion

Exclusion Criteria:

* Auto-immune disorders
* Immediate reconstruction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Grade of Radiodermatitis | During radiation treatment
  "Radiation Therapy Oncology Group" (RTOG) grading
Grade of Radiodermatitis | 90 days after radiotherapy completion
  "Radiation Therapy Oncology Group" (RTOG) grading

SECONDARY OUTCOMES:
Behavioral Risk Factor Surveillance | One day after radiotherapy completion
  Behavioral Risk Factor Surveillance System (BRFSS) Questionnaire
Behavioral Risk Factor Surveillance | 90 days after radiotherapy completion
  Behavioral Risk Factor Surveillance System (BRFSS) Questionnaire
Arm Disabilities | One day after radiotherapy completion
  Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH)
Arm Disabilities | 90 days after radiotherapy completion
  Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH)
Breast Cancer-Specific Quality of Life Questionnaire | One day after radiotherapy completion
  European Organization for Research and Treatment of Breast Cancer-Specific Quality of Life Questionnaire (EORTC QLQ-BR23)
Breast Cancer-Specific Quality of Life Questionnaire | 90 days after radiotherapy completion
  European Organization for Research and Treatment of Breast Cancer-Specific Quality of Life Questionnaire (EORTC QLQ-BR23)
Overall Quality of Life Questionnaire | One day after radiotherapy completion
  European Organization for Research and Treatment of Cancer (EORTC QLQ-30)
Overall Quality of Life Questionnaire | 90 days after radiotherapy completion
  European Organization for Research and Treatment of Cancer (EORTC QLQ-30)

CONTACTS AND LOCATIONS:
Overall Officials: Glauco Baiocchi, MD, PhD, Study Chair — AC Camargo Cancer Center
Locations (1):
- Universidade do Vale do Itajai - UNIVALI, Itajaí, Santa Catarina, Brazil